CLINICAL TRIAL: NCT03541239
Title: Immune Modulation by Ischemic Pre-conditioning in Healthy Individuals: Intracellular Signalling in Regulatory Cells
Acronym: KONDI-immun
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Fonden til Lægevidenskabens Fremme (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1-10-72-298-15
Record Dates: First submitted 2016-06-15; First posted 2018-05-30 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2016-06

CONDITIONS: Ischemia Reperfusion Injury; Ischaemia Reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- non-ischemic preconditioning (Active Comparator): The participants will have the cuff attached to the arm, however not be inflated for the 4 cycles of remote ischemic conditioning: 1 cycle is 5 minutes of inflation followed by 5 minutes of deflation. The ischemic reperfusion injury was induced by cuff inflation by the Single Cuff Tourniquet 8000 to 200 mmHg in the arm for 20 minutes followed by reperfusion for 15 minutes.
  Interventions: Device: Single Cuff Tourniquet 8000
- ischemic preconditioning (Experimental): The blood supply to the distal part of the arm will be occluded by inflation of a single cuff to 200mmHg, by the help of the Single Cuff Tourniquet 8000, for 5 minutes separated from 5 minutes of deflation, a cycle that happens 4 times in total. The ischemic reperfusion injury was induced by cuff inflation to 200 mmHg in the arm for 20 minutes followed by reperfusion for 15 minutes.
  Interventions: Device: Single Cuff Tourniquet 8000

INTERVENTIONS:
Device: Single Cuff Tourniquet 8000 — If randomized to ischemic conditioning the cuff will be inflated as stated before. If randomized to non-ischemic conditioning the cuff will not be inflated.
  Other Names: 20-54-711; 20-54-712

SUMMARY:
The aim of the study is to investigate how phosphorylation of STAT3, p38 mitogen-activated protein kinase (MAPK), extracellular signal-regulated kinase (ERK) and protein kinase B (AKT) reacts to remote ischemic conditioning (rIC) in healthy humans, which could point to mechanisms by which rIC may protect against ischemia-reperfusion injury (IRI), and if rIC affects immune reactivity.

DETAILED DESCRIPTION:
In rIC brief episodes of non-lethal ischemia and reperfusion in one vascular bed, tissue or organ, has shown to have protective effects against IRI in various organs. The protective effect of rIC seems convincing, but to date it is not clear which mechanisms give rIC its effects, and why effects are absent in some situations. Effects of rIC on the immune system are also not clear, but important if rIC is used in transplantation and autoimmunity settings, and also in regards to infection risk. Patients studied have often been given medical treatment and/or have comorbidities affecting the results.

This project will measure how intracellular phosphorylation of STAT3, p38 MAPK, ERK and AKT, inflammatory cell patterns and cytokine production react to rIC in healthy humans, and potentially give a better understanding of the mechanisms that mediate the protective effects of rIC. The intracellular mediators studied are involved in the initiation of cytokine production and regulate apoptosis and activation of the inflammatory cells. An altered balance between leucocytes and their mediators could be of importance for rIC effects, particularly in transplantation and autoimmunity, and this will be elucidated in our study.

As a secondary end point the investigators will measure the effect of rIC on pulse variability and blood pressure using a non-invasive device, since evidence regarding these aspects is sparse, although documented positive effects of rIC have primarily been on the heart and vascular system.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and well

Exclusion Criteria:

* Smoker.
* Taking regular medication.
* Any acute, chronic or systemic disease
* No hard physical exercise 72 hours prior to study participation.
* No alcohol or caffein-containing drinks 24 hours prior to study participation.
* Fasted for at least 6 hours prior to study participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2016-07-19 (Actual); Study Completion 2016-07-19 (Actual)

PRIMARY OUTCOMES:
Changes in the amount of immune cells in the peripheral blood | Baseline before any intervention, 0 minutes and 85 minutes after IRI and 24 hours after IRI
  The investigators measured the effect of ischemic preconditioning on ischemia reperfusion injury in a randomised controlled cross-over trial with healthy participants. Peripheral blood before and after the intervention was measured.
Changes in inflammatory cytokines in the peripheral blood | Baseline before any intervention, 85 minutes after IRI and 24 hours after IRI
  The investigators measured the effect of ischemic preconditioning on ischemia reperfusion injury in a randomised controlled cross-over trial with healthy participants. Peripheral blood before and after the intervention was measured.
Changes in intracellular activation markers in T-cells | Baseline before any intervention, 0 minutes and 85 mins after IRI and 24 hours after IRI
  The investigators measured the effect of ischemic preconditioning on ischemia reperfusion injury in a randomised controlled cross-over trial with healthy participants. Peripheral blood before and after the intervention was measured.
Changes in intracellular activation markers in monocytes | Baseline before any intervention, 0 minutes and 85 minutes after IRI and 24 hours after IRI
  The investigators measured the effect of ischemic preconditioning on ischemia reperfusion injury in a randomised controlled cross-over trial with healthy participants. Peripheral blood before and after the intervention was measured.

SECONDARY OUTCOMES:
Measure pulse variability. | Baseline before any intervention and until 85 minutes after IRI and 24 hours.
  Pulse variability was measured during the experiment.
Measure blood pressure. | Baseline before any intervention and until 85 minutes after IRI and 24 hours.
  Blood pressure was measured during the experiment.

CONTACTS AND LOCATIONS:
Overall Officials: Bente Jespersen, Professor, Principal Investigator — Dept. of Renal Diseases, SKS, DK; Bjarne Kuno Møller, MD, Study Chair — Dept. of Clinical Immunology, SKS, DK; Carla Baan, Professor, Study Chair — Erasmus Medical Center
Locations (1):
- C-Laboratorium, Skejby Sygehus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No